CLINICAL TRIAL: NCT06892067
Title: Safety Assessment of Over-the-counter Personal Care and Cosmetic Products Ingredients Based on Product Description and Properties
Brief Title: Safety Assessment of Over-the-counter Personal Care and Cosmetic Products Ingredients Based on Product Description
Status: Completed | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/024
Record Dates: First submitted 2024-12-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cosmetic Product Causing Toxic Effect
MeSH Terms: interventions — Cosmetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Combination Product: Cosmetic Products — To evaluate and analyze the safety of commonly used ingredients in over-the-counter personal care and cosmetic products.

SUMMARY:
"Personal care and cosmetic products maintain hygiene, enhance aesthetics and promote wellbeing. This category includes various formulations for cleansing, grooming and beautification products for skin, hair, nails, lips and teeth.

DETAILED DESCRIPTION:
This study evaluates the safety of ingredients in 100 over the counter personal care and cosmetic products. Stratified sampling selects products from various categories, brands and retailers.

ELIGIBILITY:
Inclusion Criteria:

* Over the counter personal care products available for consumer purchase,Products from various categories (e.g., skincare, haircare, makeup, eye care),
* Products from different brands and manufacturers,Products with ingredient labels or lists available,Products marketed for general consumer use (not specialized or prescription products).

Exclusion Criteria:

* Prescription-only products or those requiring medical supervision,Products intended for specialized use (e.g., medical conditions, sensitive skin)
* Products without ingredient labels or lists.
* Products from obscure or unreliable manufacturers
* Products with expired or near-expired ingredients.
* Products with unclear or misleading labelling,Products not intended for general consumer use (e.g., professional salon products),Products with ingredients already known to be harmful or banned by regulatory agencies.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Safety Assessment of Over-the-counter Personal Care and Cosmetic Products' Ingredients Based on Product Description.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Likert scales | 12 months
  Likert scales commonly comprise either five or seven options. The options on each end are called response anchors. The midpoint is often a neutral item, with positive options on one side and negative options on the other. Each item is given a score from 1 to 5 or 1 to 7

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacies (Mehmood Pharmacy, Servaid Pharmacy, Clinix+ Pharmacy), Supermarkets (Hyperstar, Metro cash and carry, Imtiaz supermarket), Departmental stores (AL Fatah, Haji cream bakhsh, Enem store), Online retailers (Saloni.pk, Just4Girls.pk, Daraz.pk), Lahore, Punjab Province, Pakistan